CLINICAL TRIAL: NCT04101812
Title: A Non-randomized, Prospective Clinical Study of Pegylated Liposomal Doxorubicin and PD-1 in the Second-line Treatment of Relapse or Metastatic Muscle Invasive Bladder Cancer
Brief Title: Pegylated Liposomal Doxorubicin, PD-1 in Treating Muscle Invasive Bladder Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Second Hospital (Other)
Collaborators: CSPC Pharmaceutical Group Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DMSMIBC-01
Record Dates: First submitted 2019-09-17; First posted 2019-09-24 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Muscle Invasive Bladder Cancer
MeSH Terms: interventions — liposomal doxorubicin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Experimental group Pegylated liposomal doxorubicin 40mg/m2 iv every 3 weeks, for 3 cycles; PD-1 every 3 weeks, for 3 cycles.
  Interventions: Drug: pegylated liposomal doxorubicin (PLD); Drug: PD-1
- Control group (Active Comparator): PD-1 every 3 weeks, for 6 cycles.
  Interventions: Drug: PD-1

INTERVENTIONS:
Drug: pegylated liposomal doxorubicin (PLD) — PLD is an anthracycline topoisomerase II inhibitor that is encapsulated in liposomes for intravenous use.
  Other Names: Doxorubicin Hydrochloride Liposome Injection
  Arms: Experimental group
Drug: PD-1 — PD-1 monoclonal antibody is a programmed death-1 (PD-1) immune checkpoint inhibitor antibody, which selectively interferes with the combination of PD-1 with its ligands and PD-L1.

SUMMARY:
Despite primary surgical management of muscle invasive bladder cancer (MIBC) with radical cystectomy and pelvic lymphnode dissection, up to 50% of patients will eventually develop tumours at distant sites, owing to pre-existing disseminated occult micrometastases. The first line treatment for relapse or metastatic MIBC is gemcitabine and cisplatin. After the failure of first line treatment, second line chemotherapy drugs can be chosen from doxorubicin, docetaxel, pemetrexed, etc. This non-randomized, prospective study aims to explore the efficacy and safety of PEGylated liposomal doxorubicin and PD-1 in second line treatment of MIBC.

ELIGIBILITY:
Inclusion Criteria:

* Clinically confirmed muscle-invasive bladder cancer.
* Histologically confirmed by HE staining or IHC staining.
* Life expectancy of greater than or equal to 3 months.
* KPS performance >60, ECOG performance status ≤2.
* Adequate liver function with a bilirubin up to 1.5 x ULN. Transaminases up to 2.5 x ULN; for liver metastasis, transaminases up to 5 x ULN.
* Adequate bone marrow function, as defined by neutrophils count of ≥1.5×109/L, platelet count≥80×109/L, hemoglobin≥9.0g/dL.
* Adequate renal function (serum creatinine ≤1.25 times the ULN, and the release rate of which ≥ 60ml/min).
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.
* Negative serum pregnancy test for female subjects with reproductive potential =< 7 days prior to registration, for women of childbearing potential only. All female patients of childbearing age and all male patients with partners of childbearing age should use a reliable method of contraception, such as the barrier method, throughout the study and for 8 weeks after last treatment.
* Sign the informed consent before any trial related activities.

Exclusion Criteria:

* A prior malignancy, other than non-melanoma skin cancer, carcinoma in situ, localized prostate cancer or ductal carcinoma in situ treated by surgery unless they have completed therapy at least 5 years prior to start of study and have no evidence of recurrent or residual disease
* Chemotherapy, biological therapy or other anti-cancer drugs ≤ 28 days prior to pre-registration
* Factors that would affect taking medicine orally, such as dysphagia, chronic diarrhea and intestinal obstruction
* History of arterial/venous thrombus ≤ 6 months prior to registration, such as cerebrovascular accident, deep vein thrombosis and pulmonary embolism
* History or tendency of gastrointestinal hemorrhage caused by severe gastroesophageal varices or other reasons.
* Dysfunction of blood coagulation: prothrombin time (PT)>16s, activated partial thromboplastin time (APTT) >43s, thrombin time (TT) >21s, INR >2, fibrinogen < 2g/L, bleeding tendency or under thrombolytic or anticoagulant therapy
* Uncontrolled intercurrent illness including, but not limited to:

ongoing or active infection; poor controlled diabetes (FBG > 10 mmol/L); urine protein ≥++, and UAE > 1.0g/24h; myocardial ischemia; congestive heart failure; cardiac arrhythmia or cardiac insufficiency; LVEF < 50%

* Unhealed wounds, ulcers or fractures
* Abuse of psychotropic substances or mentally disturbed
* History of HIV, organ transplantation or any other acquired, congenital immunodeficiency diseases
* Patients evaluated not suitable for the study in the opinion of investigators

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-09-17 (Actual); Primary Completion 2020-05-31 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Disease control rate | at least 10 months
  Disease control rate defined as confirmed complete response or partial response or stable disease under RECIST 1.0 criteria.
Objective response rate | at least 10 months
  Objective response rate defined as confirmed complete response or partial response under RECIST 1.0 criteria.

SECONDARY OUTCOMES:
Progression free survival | at least 10 months
  Progression-free survival estimated using Kaplan-Meier methods is defined as the time from registration to the earlier of death or disease progression.
Overall survival | at least 10 months
  Overall survival estimated using Kaplan-Meier methods is defined as the time from treatment initiation to death by any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical Unversity Second Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided